CLINICAL TRIAL: NCT06995417
Title: Discontinuation of Tobacco Dependence in Smoking Patients With Squamous Cell Carcinoma of the Head-neck District: Multicenter Prospective Observational Study
Acronym: STOP-HNC
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Full Professor, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: STOP-HNC
Record Dates: First submitted 2025-03-31; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cancer of Head and Neck
Keywords: Cancer Head&Neck; Smoker
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Smoking counseling — The investigator, upon enrollment, will initiate a standardized strategy from clinical practice: the investigator will conduct brief counseling ("minimal advice") using the administration of of a questionnaire that will include, in addition to questions about current and past, the administration of the Fagerstrom test to measure physical dependence on nicotine and questions to investigate intention to quit smoking (Mondor test)

SUMMARY:
The primary objective of our study is to evaluate the effectiveness of a standardized clinical practice counseling strategy for promoting post-diagnosis smoking cessation among patients with SCCHN. Efficacy will be measured as the percentage of patients who succeed in sustained smoking cessation ("sustained quitters," see below) at 6+1 months after enrollment, i.e., after the initiation of anti-smoking counseling.

ELIGIBILITY:
Inclusion criteria.

* Patients with SCCHN tumors of the oral cavity, oropharynx, hypopharynx, larynx, nasopharynx, and paranasal sinuses.
* Patients older than 18 years of age with SCCHN of these sites who are candidates for surgical/radiotherapy (RT)/radiochemotherapy (RTCT) treatment with curative intent (primary treatment).
* Patients with SCCHN who are active smokers, or have quit smoking for less than 30 days, at the time of initiation of the process (visits and instrumental tests) that led to the diagnosis of cancer

Exclusion criteria

* Patients with SCCHN cancer who have quit smoking for more than 30 days at the time of initiation of the diagnostic process.
* Patients using only e-cigarettes at the time of initiation of the treatment process.
* Patients with non-SCCHN cancer in recurrent metastatic stage and not eligible for curative purpose therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients with SCCHN who are active smokers, or have quit smoking for less than 30 days, at the time of initiation of the process (visits and instrumental examinations) that led to the cancer diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of a standardized counseling strategy in clinical practice to promote smoking cessation | 6+1 months from enrollment, i.e., initiation of anti-smoking counseling.
  The primary objective of our study is to evaluate the effectiveness of a standardized clinical practice counseling strategy for promoting post-diagnosis smoking cessation among patients with SCCHN. Efficacy will be measured as the percentage of patients who succeed in sustained smoking cessation ("sustained quitters," see below) at 6+1 months after enrollment, i.e., after the initiation of anti-smoking counseling.

CONTACTS AND LOCATIONS:
Overall Officials: LORENZO LL LIVI, MEDICAL DOCTOR, Principal Investigator — Aou Careggi
Locations (1):
- Azienda Ospedaliera Careggi, Florence, Firenze, Italy

IPD SHARING:
Plan to Share IPD: Undecided